CLINICAL TRIAL: NCT05719740
Title: Osteocrin ,a Novel Predictive Bone-derived Humoral Factor,in Diabetes Mellitus, and Its Relation With Glycemic Control and Vascular Complications
Brief Title: Osteocrin and Vascular Complications
Acronym: Osteocrin
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Walaa Soliman Hussein, principal investigator, Assiut University
Other Study IDs: Nephrologist
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-01

CONDITIONS: Whether Osteocrin Levels Are Associated With Glycemic Control, Vascular Disorders in Diabetic Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 45 patients in type 1 .DM: TYPE 1 DIABETES MELLITUS
  Interventions: Diagnostic Test: osteocrin
- and 45 patients in type 2DM: TYPE 2 DIABETES MELLITUS
  Interventions: Diagnostic Test: osteocrin

INTERVENTIONS:
Diagnostic Test: osteocrin — laboratory routine test
  Other Names: laboratory routine test

SUMMARY:
In this study, we aimed to describe the role of bone-derived factor (osteocrin) in glucose metabolism, micro and macrovascular complications in diabetic patients. Thus, further investigations of the endocrine system through bone-derived hormones may provide as new perspectives on the prediction, prevention, and treatment of diabetes mellitus.

DETAILED DESCRIPTION:
Diabetes mellitus (DM) remained the most common metabolic disorder worldwide occupying the 8th leading cause of death.[1] Defining new predictive biomarkers in diabetes would provide a window of opportunity for preventive and/or therapeutic interventions to prevent or delay the onset of irreversible long-term micro and or macro vascular complications. Progressive micro vascular vaso-degeneration is the major factor in progression of diabetic complications and contribute greatly to the increased mortality and morbidity. [2] Where Hemodynamic-mediated vascular injury was considered as one mechanism in the pathogenesis of diabetic nephropathy. [3] Bone disorders have been drawing attention as a novel diabetic complication, and diabetes is associated with an increased risk of osteoporotic fracture [4-6]. Bone is considered as an endocrine organ that influences various organs and tissues via the secretion of multiple bone derived hormones [7-8]. These endocrinal functions are, for example, glucose homeostasis [9], appetite control [10], fat deposition [11], skeletal muscle adaptation [12], male fertility [13], and cognition [14].

Therefore, these bone-derived hormones can become useful biomarkers for predicting the incidence of diabetes and the progression of diabetic complications. Osteocrin (OSTN), a bone-derived humoral factor, is a small secreted peptide cloned from bone and muscle complementary DNA (cDNA) libraries [15]. Osteocrin (Ostn) is secreted protein produced by cells of the osteoblast lineage that shows a well conserved homology with members of the natriuretic peptide (NP) family with prohormone-like characteristics [17]. To date, the exact role of Ostn has not been elucidated.

In this study, we aimed to describe the role of bone-derived factor (osteocrin) in glucose metabolism, micro and macrovascular complications in diabetic patients. Thus, further investigations of the endocrine system through bone-derived hormones may provide as new perspectives on the prediction, prevention, and treatment of diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

- Cases of the study will select randomly, based on inclusion criteria that included

* Patients were diagnosed with diabetes mellitus according to American Diabetes Association
* Age range 20-70 years
* No apparent vascular abnormalities and Acute complications

Exclusion Criteria:

* Patients are excluded for participation in the study if

  * Patients had past history of cardiovascular events (heart failure or history of coronary artery disease),
  * infections,
  * aacute diabetic complications,
  * diabetic patients on regular hemodialysis .
  * acute illness, malignancy, or pregnancy.

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: the estimated minimum required sample size is 90 patients ( 45 patients in type 1 and 45 patients in type 2).
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
to test and evaluate the role of bone-derived factor (osteocrin) in glucose metabolism,in diabetic patients with risk of micro and macrovascular complications . | 2 years

SECONDARY OUTCOMES:
to identify bone-derived factor (osteocrin) may provide as new perspectives on the prediction, prevention, and treatment of diabetes mellitus | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- walaa soliman Hussien, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided